CLINICAL TRIAL: NCT04564690
Title: Effect of Enriched QUARTET® Hen Eggs on Cardiovascular Function in Cardiovascular Patients and Healthy Individuals
Brief Title: Enriched QUARTET® Hen Eggs and Cardiovascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Head of Scientific center of excellence for personalized health care, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #KK.01.1.1.01.0010
Record Dates: First submitted 2020-07-02; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: n-3 Polyunsaturated Fatty Acids; Selenium; Vitamin E; Lutein
Keywords: n-3 polyunsaturated fatty acids; selenium; vitamin E; lutein; vascular function; endothelium; cardiovascular health
MeSH Terms: interventions — Fatty Acids, Omega-3; Selenium; Vitamin E; Lutein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QUARTET® (Experimental): Consumption of three QUARTET® (n-3 PUFA, selenium, vitamin E, lutein enriched) hen eggs per day for three weeks
  Interventions: Dietary Supplement: QUARTET® hen eggs (enriched in n-3 PUFA, selenium, vitamin E and lutein)
- Control (Experimental): Consumption of three regular hen eggs per day for three weeks
  Interventions: Dietary Supplement: Regular hen eggs

INTERVENTIONS:
Dietary Supplement: QUARTET® hen eggs (enriched in n-3 PUFA, selenium, vitamin E and lutein) — Consumption of three QUARTET® hen eggs (enriched in n-3 PUFA, selenium, vitamin E and lutein) per day for three weeks
  Arms: QUARTET®
Dietary Supplement: Regular hen eggs — Consumption of three regular hen eggs per day for three weeks
  Arms: Control

SUMMARY:
Role of oxidative stress in the development of cardiovascular diseases is well known and extensively investigated, because of its direct effects on vascular function, but also on the activation of the immune response. Thus, food products that could increase the antioxidant capacity of the vascular system would also act protective against cardiovascular diseases. However, we lack systematic clinical and pre-clinical research with food products instead of food supplements, which would result in consistent and repeatable results. Many studies have proven the effectiveness of n-3 polyunsaturated fatty acids (n-3 PUFA) in improvement of endothelial function, improvement of elasticity of the vascular wall and the anti-inflammatory effects in patients with chronic diseases, such as metabolic syndrome, if they are taken as an pharmacological preparation. Our research group recently reported that favorable anti-inflammatory properties of n-3 PUFA enriched hen eggs potentially contribute to the improvement of microvascular endothelium-dependent vasodilation in healthy individuals. In addition, this study aimed to determine the effect of QUARTET® hen eggs (enriched in n-3 PUFA, selenium, vitamin E and lutein; QUARTET No. 012743696, 2014.) consumption on cardiovascular function in both healthy individuals and cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (sedentary)
* healthy volunteers (athletes)
* cardiac patients (patients with acute myocardial infarction, hypertensive patients with/without hypertensive heart disease, heart failure patients)

Exclusion Criteria for Healthy Volunteers:

* oral contraceptives
* drugs that could affect endothelium
* hypertension
* coronary artery disease
* diabetes
* hyperlipidaemia
* renal impairment
* cerebrovascular and peripheral artery disease

Exclusion Criteria for Cardiac Patients:

* known malignant disease
* hereditary metabolic diseases and other hereditary systemic diseases
* autoimmune diseases or systemic diseases with immunopathology
* unregulated hypertension
* recent surgery (3 months)
* recent significant trauma (6 months)
* renal insufficiency (except in diabetic patients unless Endogenous Creatinine Clearance > 60ml / min)
* active bleeding (hematuria, GI tract, menorrhagia)
* fresh ICV (6 weeks)
* neurodegenerative diseases and epilepsy
* significant anemia (Hg <110 (men), <100 (women))
* condition after resuscitation (3 months)
* therapy that significantly affects vascular or immune function (monoclonal antibodies, immunosuppressants, systemic corticosteroids ...)
* chronic respiratory failure and conditions of chronic hypoxemia
* sepsis and chronic active infections with systemic inflammatory response (active tuberculosis, etc.)
* untreated thyroid disease
* active abuse of alcohol and drugs
* liver failure (advanced liver disease with impaired synthetic and metabolic function)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Microvascular reactivity | 3 weeks
  Forearm skin microvascular reactivity in response to: vascular occlusion (post-occlusion reactive hyperemia, PORH); iontophoresis of acetylcholine (endothelium-dependent) and sodium nitroprusside (endothelium-independent); and local thermal hyperemia (LTH, NO-dependent vasodilation), measured by laser Doppler flowmetry (LDF)
Macrovascular reactivity - FMD of brachial artery | 3 weeks
  Flow mediated dilation (FMD) of brachial artery measured by ultrasound.
Macrovascular reactivity - TCD of cerebral blood vessels | 3 weeks
  Vascular reactivity of cerebral blood vessels measured by transcranial Doppler (TCD).
Oxidative stress - thiobarbituric acid reactive substances (TBARS) | 3 weeks
  Measurement of biomarkers of oxidative stress level. Thiobarbituric acid reactive substances (TBARS) - biomarker of lipid peroxidation.
Oxidative stress - ferric-reducing ability of plasma (FRAP) | 3 weeks
  Measurement of biomarkers of oxidative stress level. Ferric-reducing ability of plasma (FRAP) - biomarker of plasma antioxidant capacity.
Oxidative stress - antioxidative enzymes | 3 weeks
  Measurement of biomarkers of oxidative stress level. Plasma concentration of antioxidative enzymes.
T helper lymphocyte differentiation | 3 weeks
  Regulatory T cells (Treg, Foxp3) and Th17 cells will be determined measuring intracellular expression for distinct Th17 markers by using FACS Canto II flow cytometer system.
Serum Pro- and Anti-Inflammatory Cytokines, Chemokines, Growth Factors and Soluble Cell Adhesion Molecules Protein Concentration | 3 weeks
  Measurement of serum protein concentration (pg/mL) of various pro- and anti-inflammatory cytokines, chemokines, growth factors and soluble cell adhesion molecules by kits and panels for multiplex protein quantitation using the Luminex 200 instrument platform.
Endothelial cell activation | 3 weeks
  Measurement of serum protein concentration of cell adhesion molecules (e.g. intercellular adhesion molecule 1 - ICAM-1, vascular cell adhesion protein 1 - VCAM-1, and E-selectin) by commercially available ELISA kits, or by multiplex assay kits for the Luminex platform (Luminex® 100/200™ System).

SECONDARY OUTCOMES:
Blood pressure | 3 weeks
  Measurement of systolic and diastolic blood pressure.
Serum lipid profile | 3 weeks
  Total cholesterol, triglycerides, LDL cholesterol, HDL cholesterol
Body composition | 3 weeks
  Body composition and body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Fat Free Mass (FFM kg) and Fat (Fat Mass kg).
Body fluid status | 3 weeks
  Body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Total Body Water (TBW L), Extracellular Water (ECW L), Intracellular Water (ICW L), Plasma Fluid (PF L) and Interstitial Fluid (IF L) and Body Density (kg/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Center of Excellence for Personalized Health Care, Josip Juraj Strossayer University of Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stupin A, Rasic L, Matic A, Stupin M, Kralik Z, Kralik G, Grcevic M, Drenjancevic I. Omega-3 polyunsaturated fatty acids-enriched hen eggs consumption enhances microvascular reactivity in young healthy individuals. Appl Physiol Nutr Metab. 2018 Oct;43(10):988-995. doi: 10.1139/apnm-2017-0735. Epub 2018 Apr 10. PMID 29633621
- [Background] Stupin M, Kibel A, Stupin A, Selthofer-Relatic K, Matic A, Mihalj M, Mihaljevic Z, Jukic I, Drenjancevic I. The Physiological Effect of n-3 Polyunsaturated Fatty Acids (n-3 PUFAs) Intake and Exercise on Hemorheology, Microvascular Function, and Physical Performance in Health and Cardiovascular Diseases; Is There an Interaction of Exercise and Dietary n-3 PUFA Intake? Front Physiol. 2019 Aug 30;10:1129. doi: 10.3389/fphys.2019.01129. eCollection 2019. PMID 31543828
- [Background] Stupin A, Mihalj M, Kolobaric N, Susnjara P, Kolar L, Mihaljevic Z, Matic A, Stupin M, Jukic I, Kralik Z, Grcevic M, Kralik G, Seric V, Drenjancevic I. Anti-Inflammatory Potential of n-3 Polyunsaturated Fatty Acids Enriched Hen Eggs Consumption in Improving Microvascular Endothelial Function of Healthy Individuals-Clinical Trial. Int J Mol Sci. 2020 Jun 10;21(11):4149. doi: 10.3390/ijms21114149. PMID 32532035
- [Derived] Susnjara P, Kolobaric N, Matic A, Mihaljevic Z, Stupin A, Marczi S, Drenjancevic I. Consumption of Hen Eggs Enriched with n-3 Polyunsaturated Fatty Acids, Selenium, Vitamin E and Lutein Incites Anti-Inflammatory Conditions in Young, Healthy Participants - A Randomized Study. Front Biosci (Landmark Ed). 2022 Dec 27;27(12):332. doi: 10.31083/j.fbl2712332. PMID 36624951